CLINICAL TRIAL: NCT00066365
Title: A Phase II Study of Aerosolized GM-CSF (NSC# 613795, IND# 11042) in Patients With First Pulmonary Recurrence of Osteosarcoma
Brief Title: Inhaled Sargramostim in Treating Patients With First Pulmonary (Lung) Recurrence of Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOST0221; CDR0000315540 (Other: Clinical Trials.gov); COG-AOST0221 (Other: Children's Oncology Group); NCI-2012-02543 (Other: NCI); U10CA098543 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Cancer; Sarcoma
Keywords: metastatic osteosarcoma; recurrent osteosarcoma; lung metastases
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma; Osteosarcoma | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (unilateral recurrence) - Sargramostim and thoractomy (Experimental): Patients receive initial inhalation therapy inhaled sargramostim (GM-CSF) twice daily on days 1-7. Treatment repeats every other week every 14 days for a total of 2 courses. Patients undergo surgical procedure thoracotomy on day 22. Beginning on day 29, or as soon as possible thereafter, patients begin post-thoracotomy inhalation therapy for up to 12 additional courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.
  Interventions: Biological: sargramostim; Procedure: conventional surgery
- Group 2 (bilateral recurrence) - Sargramostim and thoractomy (Experimental): Patients may be enrolled on study either before or after the first thoracotomy procedure. For the first thoracotomy, patients undergo surgical procedure unilateral thoracotomy. Patients receive initial inhalation therapy inhaled GM-CSF, as soon as possible after recovery from first thoracotomy, twice daily on days 1-7. Treatment repeats every other week every 14 days for a total of 2 courses. Patients undergo surgical procedure contralateral thoracotomy on day 22. Beginning on day 29, or as soon as possible, patients begin post-thoracotomy inhalation therapy as above for up to 12 additional courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.
  Interventions: Biological: sargramostim; Procedure: conventional surgery

INTERVENTIONS:
Biological: sargramostim — given by inhalation, dosage escalation Level 1 Dose: 240 micrograms, Level 2 Dose: 1,000 micrograms, and Level 3 Dose: 1,750 micrograms.
  Other Names: aerosol sargramostim; inhaled GM-CSF; Granulocyte Macrophage Colony Stimulating Factor; rhu GM-CSF; rGM-CSF; GM-CSF; Prokine®; Leukine®; Interberin®; NSC#613795
Procedure: conventional surgery — thoracotomy

SUMMARY:
RATIONALE: Inhaling aerosolized sargramostim before and after surgery may interfere with the growth of tumor cells and shrink the tumor so that it can be removed during surgery. Sargramostim may then kill any tumor cells remaining after surgery. This may be an effective treatment for osteosarcoma that has spread to the lung.

PURPOSE: This phase II trial is studying how well inhaled sargramostim works in treating patients who are undergoing surgery for the first recurrence of osteosarcoma that has spread to the lung.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the histological findings from patients with first pulmonary recurrence of osteosarcoma who undergo resection of pulmonary metastases after treatment with 2 courses of aerosolized sargramostim (GM-CSF).
* Determine the event-free survival of patients treated with this drug.
* Determine whether the maximum tolerated dose in the trial of inhaled GM-CSF in adult patients with melanoma is tolerable in pediatric patients.

Secondary

* Determine the effect of specific thoracic surgical management on outcome in patients treated with this drug.

OUTLINE: This is a multicenter, dose escalation study. Patients are assigned to 1 of 2 groups according to the extent of pulmonary recurrence (unilateral or bilateral).

* Group I (unilateral recurrence):

  * Initial inhalation therapy: Patients receive inhaled sargramostim (GM-CSF) twice daily on days 1-7. Treatment repeats every other week every 14 days for a total of 2 courses.
  * Thoracotomy: Patients undergo thoracotomy on day 22.
  * Post-thoracotomy inhalation therapy: Beginning on day 29, or as soon as possible thereafter, patients resume inhalation therapy as above for up to 12 additional courses.
* Group II (bilateral recurrence): Patients may be enrolled on study either before or after the first thoracotomy.

  * First thoracotomy: Patients undergo unilateral thoracotomy.
  * Initial inhalation therapy: Patients receive inhaled GM-CSF, as soon as possible after recovery from first thoracotomy, twice daily on days 1-7. Treatment repeats every other week every 14 days for a total of 2 courses.
  * Contralateral thoracotomy: Patients undergo contralateral thoracotomy on day 22.
  * Post-thoracotomy inhalation therapy: Beginning on day 29, or as soon as possible, patients resume inhalation therapy as above for up to 12 additional courses.

Treatment in both groups continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 1.6-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed osteosarcoma at primary diagnosis

  * Lesions detected in at least 1 lung that are consistent with metastatic disease and approachable with thoracotomy
  * No prior recurrence of osteosarcoma
  * No other sites of metastases
* Resectable pulmonary nodule(s), defined as nodule(s) that are removable without performing a pneumonectomy (e.g., nodules immediately adjacent to the main stem bronchus or main pulmonary vessels)
* Prior thoracotomy allowed in patients with imaging consistent with metastatic involvement in both lungs provided the lung on which the thoracotomy was performed is disease-free
* No pleural effusion or pleural based nodules

PATIENT CHARACTERISTICS:

Age

* 39 and under

Performance status

* Karnofsky 50-100% (patients over 16 years of age)
* Lansky 50-100% (patients 16 years of age and under)

Life expectancy

* At least 8 weeks

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry at least 94%
* Baseline Forced expiratory volume in 1 second (FEV_1) at least 80% of predicted
* No history of asthma
* No history of reactive airway disease
* No history of bronchospasm

Other

* Willing and able to perform inhalation therapy
* No medical contraindication to surgical excision
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy
* No other concurrent immunomodulating agents

Chemotherapy

* No concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent steroids by any route

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No concurrent thoracoscopy or video-assisted thoracic surgery

Other

* No more than 1 prior treatment regimen for osteosarcoma
* No concurrent participation in another COG therapeutic study

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2004-07; Primary Completion 2010-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carola A. Arndt, MD, Study Chair — Mayo Clinic
Locations (93):
- United States (83):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (7):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Result] Arndt CA, Koshkina NV, Inwards CY, Hawkins DS, Krailo MD, Villaluna D, Anderson PM, Goorin AM, Blakely ML, Bernstein M, Bell SA, Ray K, Grendahl DC, Marina N, Kleinerman ES. Inhaled granulocyte-macrophage colony stimulating factor for first pulmonary recurrence of osteosarcoma: effects on disease-free survival and immunomodulation. a report from the Children's Oncology Group. Clin Cancer Res. 2010 Aug 1;16(15):4024-30. doi: 10.1158/1078-0432.CCR-10-0662. Epub 2010 Jun 24. PMID 20576718

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy: Patients may be enrolled on study either before or after the first thoracotomy procedure. For the first thoracotomy, patients undergo unilateral thoracotomy. Patients receive initial inhalation therapy inhaled GM-CSF, as soon as possible after recovery from first thoracotomy, twice daily on days 1-7. Treatment repeats every other week every 14 days for a total of 2 courses. Patients undergo contralateral thoracotomy on day 22. Beginning on day 29, or as soon as possible, patients begin post-thoracotomy inhalation therapy as above for up to 12 additional courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.
  sargramostim: given by inhalation, dosage escalation Level 1 Dose: 240 micrograms, Level 2 Dose: 1,000 micrograms, and Level 3 Dose: 1,750 micrograms.
  conventional surgery: thoracotomy
Period: Overall Study
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Started | 31 | 18
Completed | 8 | 4
Not Completed | 23 | 14
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 15 | 12
Not completed — Physician Decision | 1 | 0
Not completed — No viable tumor after 1 cycle of therapy | 2 | 0
Not completed — Ineligible | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy | Total
Number analyzed (Participants) | 31 | 18 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 14 | 39
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [7 to 29] | 17 [14 to 20] | 16 [7 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 5 | 20
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 29 | 15 | 44
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 22 | 16 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 18 | 48
  Canada | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Status of FAS Ligand in Pre-chemotherapy Sample
Description: FAS ligand (FASL) is a homotrimeric type II transmembrane protein expressed on cytotoxic T lymphocytes. The Cluster of Differentiation 1a (CD1a) status is measured in Immunohistochemistry (IHC) categories.
Time Frame: 29 days after start of protocol therapy
Population: Patients who were enrolled in the unilateral recurrence group do not contribute to the assessment of any "Pre Chemotherapy" analysis. Such patients only had tissue for assessment after the first thoracotomy which was planned for 22 days after the start of sargramostim treatment. 14 patients were evaluated for this primary outcome measure.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 0 | 14
participants
  IHC Category 0 |  | 7
  IHC Category 1 |  | 5
  IHC Category 2 |  | 1
  IHC Category 3 |  | 1

2. Primary Outcome: Presence of FAS in Pre-chemotherapy Sample
Description: FAS/APO-1 is a transmembrane receptor. The presence is measured in Immunohistochemistry (IHC) categories.
Time Frame: 29 days after start of protocol therapy
Population: Patients who were enrolled in Group 1 (unilateral recurrence) do not contribute to the assessment of any "Pre Chemotherapy" analysis. Such patients only had tissue for assessment after the first thoracotomy which was planned for 22 days after the start of sargramostim treatment.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 0 | 14
participants
  IHC Category 0 |  | 5
  IHC Category 1 |  | 5
  IHC Category 2 |  | 2
  IHC Category 3 |  | 2

3. Primary Outcome: FAS Ligand in Post Chemotherapy Sample
Description: FAS ligand or FASL is a homotrimeric type II transmembrane protein expressed on cytotoxic T lymphocytes. The presence is measured in Immunohistochemistry (IHC) categories.
Time Frame: 29 days after start of protocol therapy
Population: 22 patients from the unilateral recurrence group and 13 patients from the bilateral recurrence group were evaluated for this outcome measure.
Measure: Number; unit: participants
Groups:
- Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy: Patients may be enrolled on study either before or after the first thoracotomy procedure. For the first thoracotomy, patients undergo unilateral thoracotomy. Patients receive initial inhalation therapy inhaled GM-CSF, as soon as possible after recovery from first thoracotomy, twice daily on days 1-7. Treatment repeats every other week every 14 days for a total of 2 courses. Patients undergo contralateral thoracotomy on day 22. Beginning on day 29, or as soon as possible, patients begin post-thoracotomy inhalation therapy as above for up to 12 additional courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.
  sargramostim: given by inhalation, dosage escalation Level 1 Dose: 240 micrograms, Level 2 Dose: 1,000 micrograms, and Level 3 Dose: 1,750 micrograms
  conventional surgery: thoracotomy
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 22 | 13
participants
  IHC Category 0 | 16 | 7
  IHC Category 1 | 4 | 2
  IHC Category 2 | 1 | 2
  IHC Category 3 | 1 | 2

4. Primary Outcome: FAS Status in Post Chemotherapy Sample
Description: FAS/APO-1 is a transmembrane receptor. The presence is measured in Immunohistochemistry (IHC) categories.
Time Frame: 29 days after start of protocol therapy
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 22 | 13
participants
  IHC Category 0 | 14 | 5
  IHC Category 1 | 4 | 4
  IHC Category 2 | 1 | 0
  IHC Category 3 | 3 | 4

5. Primary Outcome: CD1a Status in Pre Chemotherapy Sample
Description: CD1a (Cluster of Differentiation 1a) is a human protein encoded by the CD1A gene, presence is measured by positivity.
Time Frame: 29 days after start of protocol therapy
Population: Patients enrolled in the unilateral recurrence group do not contribute to the assessment of any "Pre Chemotherapy" analysis. Such patients only had tissue for assessment after the first thoracotomy which was planned for 22 days after the start of sargramostim treatment. 7 patients were evaluated from the bilateral recurrence group.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 0 | 7
participants
  Negative |  | 5
  Focally Positive |  | 2

6. Primary Outcome: CD1a Status in Post Chemotherapy Sample
Description: CD1a (Cluster of Differentiation 1a) is a human protein encoded by the CD1A gene, presence is measured by positivity.
Time Frame: 29 days after start of protocol therapy
Population: 20 patients were evaluated for this outcome measure from the unilateral group and 7 patients were evaluated from the bilateral group.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 20 | 7
participants
  Negative | 8 | 5
  Focally Positive | 12 | 2

7. Primary Outcome: S100 Status in Pre Chemotherapy Sample
Description: The S-100 proteins are a family of low-molecular-weight proteins characterized by two calcium-binding sites that have helix-loop-helix ("EF-hand type") conformation.
Time Frame: 29 days after start of protocol therapy
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 0 | 7
participants
  Negative |  | 4
  Focally Positive |  | 3

8. Primary Outcome: S100 Status in Post Chemotherapy Sample
Description: as for outcome 7
Time Frame: 29 days after start of protocol therapy
Population: 20 patients from the unilateral recurrence group and 10 patients from the bilateral recurrence group were evaluated for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 20 | 10
participants
  Negative | 17 | 9
  Focally Positive | 3 | 1

9. Primary Outcome: Clusterin Status in Pre Chemotherapy Sample
Description: The protein encoded by this gene can under some stress conditions also be found in the cell cytosol. It has been suggested to be involved in several basic biological events such as cell death, tumor progression, and neurodegenerative disorders.
Time Frame: 29 days after start of protocol therapy
Population: Patients enrolled in the unilateral recurrence group do not contribute to the assessment of any "Pre Chemotherapy" analysis. Such patients only had tissue for assessment after the first thoracotomy which was planned for 22 days after the start of sargramostim treatment. 7 patients were measured from the bilateral recurrence group.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 0 | 7
participants
  Negative |  | 5
  Focally Positive |  | 2

10. Primary Outcome: Clusterin Status in Post Chemotherapy Sample
Time Frame: 29 days after start of protocol therapy
Population: This outcome measure was evaluated in 30 patients, 20 patients in the unilateral recurrence group and 10 patients in bilateral recurrence group.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 20 | 10
participants
  Negative | 17 | 7
  Focally Positive | 3 | 3

11. Primary Outcome: Event Free Survival (EFS)
Description: EFS defined as the time from enrollment on the study until disease progression, occurrence of a second malignant neoplasm (SMN), death or last contact, whichever comes first. Disease progression, occurrence of a SMN or death will be considered an analytic even. In all other cases, the patient will be considered censored at last contact.
Time Frame: Time of enrollment to Event or 5 years from enrollment, whichever occurs first
Population: There were 4 ineligible unilateral patients and 2 ineligible bilateral patients not included in this analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 27 | 16
years | .57 [.31 to .68] | .33 [.19 to .49]

12. Primary Outcome: Feasibility Success
Description: Feasibility success defined as received 21 days of protocol therapy, did not experience grade III or grade IV toxicity according to Common Toxicity Criteria for Adverse Events (CTCAE) version 3 and rendered surgically free of disease in the lungs.
Time Frame: Enrollment through 21 days of protocol therapy
Population: This outcome measure was calculated for eligible patients only. This yields 27 patients for assessment of this measure in Group 1 and 16 patients for assessment of this measure in Group 2.
Measure: Number; unit: participants
Arm/Group | Group 1 (Unilateral Recurrence) - Sargramostim and Thoractomy | Group 2 (Bilateral Recurrence) - Sargramostim and Thoractomy
Number analyzed (Participants) | 27 | 16
participants
  Yes | 24 | 16
  No | 3 | 0

ADVERSE EVENTS:
Description: SAE field contains NCI Common Toxicity Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. AE counts only based on eligible patients
Groups:
- Group 1 (Unilateral Recurrence); Group 2 (Bilateral Recurrence): (See Detailed Description and Interventions for drugs, dosages, delivery method and frequency.)
  sargramostim: given by inhalation
  conventional surgery: thoracotomy
Arm/Group | Group 1 (Unilateral Recurrence) | Group 2 (Bilateral Recurrence)
Serious Adverse Events (participants affected / at risk) | 4/27 | 0/16
Other Adverse Events (participants affected / at risk) | 8/27 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Unilateral Recurrence) (N=27) | Group 2 (Bilateral Recurrence) (N=16)
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Unilateral Recurrence) (N=27) | Group 2 (Bilateral Recurrence) (N=16)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Forced expiratory volume decreased (Investigations) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Pain (General disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Vital capacity abnormal (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.